CLINICAL TRIAL: NCT01485107
Title: Feasibility Study: Evaluation of the Ulthera® System for Lifting and Tightening of the Décolleté
Brief Title: Feasibility Study: Evaluation of the Ulthera® System for Treatment of the Décolleté
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-105
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Skin Laxity of the décolleté
Keywords: Ulthera® System; Ultherapy™ treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy™ treatment on the décolleté (Experimental): All enrolled subjects will receive the study treatment.
  Interventions: Device: Ulthera® System

INTERVENTIONS:
Device: Ulthera® System — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ultherapy™ treatment

SUMMARY:
Up to 20 subjects will be enrolled. Subjects will receive treatment of the décolleté using the Ulthera® System. Subjects will be return for follow-up visits at 90 and 180 days post-treatment. The study will evaluate the effectiveness of the Ulthera® System to lift and tighten the skin of the décolleté region.

DETAILED DESCRIPTION:
This is a prospective, single-center study. Baseline Fabi/Bolton 5-Point Chest Wrinkle scale scores and chest measurements will be assessed prior to study treatment. Study images will be obtained pre-treatment, immediate post-treatment, and at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 35 to 60 years.
* Subject in good health.
* Moderate to severe (grade of ≥3 on Fabi/Bolton scale) skin laxity on the décolleté.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Scarring in areas to be treated.
* Tattoos in the areas to be treated.
* Patients with ports or defibrillators.
* Breast size >400cc each as measured by water displacement method.
* History of breast reduction surgery.
* Any open wounds or lesions in the area.
* Active and severe inflammatory acne in the region to be treated.
* Patients who have a history with keloid formation or hypertropic scarring

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Improvement in overall lifting and tightening of skin | 90 days post-treatment
  Lifting and tightening of décolleté skin as determined by a masked, qualitative assessment of photographs at 90 days posttreatment compared to baseline.

SECONDARY OUTCOMES:
Skin Laxity of the Décolleté | 90 and 180 days post-treatment
  The amount of skin laxity will be assessed using the Fabi/Bolton 5-Point Chest Wrinkle Scale. Skin laxity will be assessed at each follow-up visit compared to baseline.
Bilateral chest measurements | 90 and 180 days post-treatment
  Measurements from mid-clavicle to nipple obtained at each follow-up visit compared to baseline to assess for lifting and tightening of skin.
Overall aesthetic improvement | 90 and 180 days post-treatment
  Based on Global Aesthetic Improvement Scale (GAIS) scores.
Patient satisfaction | 90 and 180 days post-treatment
  Subject-completed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldman, MD, Principal Investigator — Goldman, Butterwick, Fitzpatrick & Groff of Dermatology Cosmetic Laser
Locations (1):
- Goldman, Butterwick, Fitzpatrick & Groff of Dermatology Cosmetic Laser, San Diego, California, United States